CLINICAL TRIAL: NCT00479791
Title: Lipid, Glycemic, and Insulin Responses to Meals Rich in Saturated, Cis-Monounsaturated, and Polyunsaturated Fatty (n-3 and n-6)Acids in Subjects With Type 2 Diabetes Mellitus
Brief Title: Lipid, Glycemic, and Insulin Responses to Meals Rich in Different Fatty Acids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: M01RR000633 (NIH)
Record Dates: First submitted 2007-05-24; First posted 2007-05-28 (Estimated); Last update posted 2007-05-28 (Estimated); Status verified 2007-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes mellitus; Fatty acids; Postprandial response; Insulin; Glucose; Triglycerides
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Test meals rich in different fatty acids

SUMMARY:
A meal rich in very-long chain omega-3 fatty acids or oleic acid may lower postprandial insulin levels in comparison to a meal rich in linoleic acid or palmitic acid. A meal rich in very long-chain omega-3 fatty acids may lower postprandial triglyceride levels compared to other fatty acids.

DETAILED DESCRIPTION:
Research Design and Methods: Test meals rich in palmitic acid, linoleic acid, oleic acid, and eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA) and containing 1,000 kcal each were administered in a randomized cross-over design every 3 to 4 days to 11 patients with T2DM. Serum insulin, glucose, and triglycerides concentrations were measured for 360 minutes. All subjects received an isoenergic diet of constant composition throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus not on insulin therapy

Exclusion Criteria:

* Thyroid, renal, or hepatic disease, uncontrolled hypertension, anemia, history of ketosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 1997-04; Study Completion 1999-06 (Actual)

PRIMARY OUTCOMES:
Insulin, and glucose | 15 days

SECONDARY OUTCOMES:
Triglycerides | 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Abhimanyu Garg, MD, Study Chair — UT Southwestern Medical Center at Dallas
Locations (1):
- UT Southwestern Medical Center at Dallas, Dallas, Texas, United States